CLINICAL TRIAL: NCT06528119
Title: The Combined Usage of Clinical Physical Finding With Simple Triage and Rapid Treatment (START), Modified Early Warning Score(MEWS)and Quick Sequential Organ Failure Assessment(qSOFA) in Management of COVID 19 Patients
Brief Title: The Combined Usage of Clinical Physical Finding in Management of COVID 19 Patients
Status: Completed | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, Physician of Emergency Medicine, St. Martin De Porress Hospital
Other Study IDs: 22B-005
Record Dates: First submitted 2024-07-29; First posted 2024-07-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Pandemic
Keywords: blood pressure; heart rate; respiratory rate; consciousness status; quick Sequential Organ Failure Assessment (qSOFA)
MeSH Terms: conditions — COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID 19 pandemic — Physiological indicators such as blood pressure, heart rate, respiratory rate, and consciousness status of COVID-19 patients are used to apply the START, MEWS, and qSOFA in COVID-19 patients.(COVID 19 病患).

SUMMARY:
Physiological indicators such as blood pressure, heart rate, respiratory rate, and consciousness status of COVID-19 patients are used to apply the START (simple triage and rapid treatment, START), Modified Early Warning Score (MEWS), and quick Sequential Organ Failure Assessment (qSOFA) as tools for assessing clinical symptom tracking, deterioration, and subsequent improvement in COVID-19 patients. In response to the need for scarce manpower when a large number of emergency patients appear, a simple and easy-to-operate assessment method is adopted for mild patients, and artificial intelligence technology can be further used to assist in the assessment for early response and medication.

DETAILED DESCRIPTION:
Due to the development of the pandemic , the virus has constantly mutated, leading to a vast majority of mild cases. This has significantly increased the burden on medical personnel. The investigators are trying to find a way to track whether their clinical symptoms have worsened. At the same time, the investigators want to know the changes in patient symptoms in real-time through online monitoring This is a single-center retrospective study of a group of COVID-19 patients. Review their medical records, mainly based on hospital field records and existing physiological indicators of patients such as blood pressure, heart rate, respiratory rate, and consciousness status. The partients visited the hospital between March 2020 and September 2022. All patients were given physiological value indicators MEWS, qSOFA, and START for scoring and assess the clinical symptom deterioration of COVID-19 patients.

In this study, The investigators collect the physiological values of each patient and the data on the nursing records during hospitalization to judge whether the symptoms have worsened

ELIGIBILITY:
Inclusion Criteria:

* a group of hospitalized COVID 19 patients were treated in the hospital between March 2020 and Sep.2022

Exclusion Criteria: Exclude patients who lack information in their medical records and incomplete clinical data.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID 19 patients were treated in the hospital between March 2020 and Sep.2022
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
COVID 19 pandemic | March 2020 and September 2022
  Assessing clinical symptom tracking, deterioration, and subsequent improvement in COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsi Chen, MD, Principal Investigator — St. Martin De Porres Hospital,emergency medicine
Locations (1):
- St. Martin De Porres Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No